CLINICAL TRIAL: NCT02346409
Title: Cerebello-thalamo-cortical Coupling in Essential Tremor: Effects of High Frequency tACS of the Cerebellum
Brief Title: Cerebello-thalamo-cortical Coupling in Essential Tremor
Acronym: CERESTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C14-44; 2014-A01393-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2015-01-05; First posted 2015-01-27 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2021-08

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LFP-MEG recording with tACS of the cerebellum (Experimental): To explore how cerebellar stimulation (using tACS) will alter oscillations and coupling along the CTC pathway, relating these changes in brain activity to clinical improvement.
  Interventions: Device: tACS of the cerebellum
- tACS of the cerebellum vs VIM-DBS (Active Comparator): To evaluate the differential effects of non invasive high-frequency stimulation tACS of the cerebellum, as compared to high-frequency stimulation of the thalamus (using DBS of the VIM).
  Interventions: Device: tACS of the cerebellum

INTERVENTIONS:
Device: tACS of the cerebellum — tACS of the cerebellum

SUMMARY:
Essential tremor (ET) is a frequent and disabling disorder with progressive worsening of postural tremor of the upper limbs that impairs most of the manual activities of every day life (feeding, drinking, etc.). Although the pathophysiology of essential tremor (ET) is not fully elucidated, tremor is associated with abnormal activity within different brain regions, in particular the thalamus and the cerebellum. Deep brain stimulation (DBS) of the ventral intermediate nucleus of the thalamus (VIM-Thal) reverses the symptoms of tremor but is an invasive procedure. Transcranial stimulation of the cerebellum may represent a non-invasive therapeutic option for ET patients. Here, the investigators propose to test the efficacy of cerebellar stimulation in 15 ET patients previously operated for DBS of the thalamus. To further understand how this treatment provokes tremor reduction, the investigators will analyse the brain neuronal activity in 13 others ET patients candidate to thalamic DBS by using combined electrophysiological recordings of the thalamus (with the electrodes implanted), the cerebellum and the cortex with magnetoencephalography.

ELIGIBILITY:
Inclusion Criteria:

* age below 75 years
* diagnosis of essential tremor according to the criteria of the Tremor Investigation Group and the Consensus statement of the Movement Disorder Society Group (ref)
* health insurance
* signed informed written consent

Exclusion Criteria:

* other neurological disorders
* medications that interact with or influence brain excitability
* significant brain lesions detected in MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
The neuronal activity in the cerebello-thalamo-cortical pathway | 1 day
  LFP, MEG and EMG activity recordings

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olivier C, Lamy JC, Kosutzka Z, Van Hamme A, Cherif S, Lau B, Vidailhet M, Karachi C, Welter ML. Cerebellar Transcranial Alternating Current Stimulation in Essential Tremor Patients with Thalamic Stimulation: A Proof-of-Concept Study. Neurotherapeutics. 2023 Jul;20(4):1109-1119. doi: 10.1007/s13311-023-01372-6. Epub 2023 Apr 25. PMID 37097344